CLINICAL TRIAL: NCT05385055
Title: A Cross-sectional, Multi-regional Study to Demonstrate Reduction in Exposure to Key Toxicants, Oxidative Stress, and Inflammation Following At Least 2 Years of Tobacco Heating System (THS) Use Compared to Cigarette Smoking
Brief Title: Reduction of Exposure, Inflammation, and Oxidative Stress Following At Least 2 Years of Switching to THS Use Compared to Cigarette Smoking
Status: Completed | Type: Observational
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: P1-RMC-03-INT
Record Dates: First submitted 2022-05-17; First posted 2022-05-23 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Inflammation; Oxidative Stress; Smoking; Smoking Abstinence
MeSH Terms: conditions — Inflammation; Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cigarette: Current cigarette smokers
  Interventions: Other: Cigarette smoking
- THS: THS users with a minimum of 2 years of THS use
  Interventions: Other: THS use
- SA: Former cigarette smokers with minimum of 2 years of smoking abstinence
  Interventions: Other: Smoking abstinence

INTERVENTIONS:
Other: THS use — N/A: No intervention was assigned.
  Groups: THS
Other: Cigarette smoking — N/A: No intervention was assigned.
  Groups: Cigarette
Other: Smoking abstinence — N/A: No intervention was assigned.
  Groups: SA

SUMMARY:
This is a cross-sectional 3-group study with subjects enrolled and matched by region (Asia, Europe), age, sex, and average daily product consumption over the last 2 years as self-reported. The study will be conducted as a multi-center and multi-regional study, to demonstrate beneficial effects of switching from cigarettes to THS.

DETAILED DESCRIPTION:
The purpose of this study is primarily to demonstrate beneficial effects of switching from cigarette smoking to THS use for at least 2 years compared to cigarette smoking in a real-life condition on both inflammation and oxidative stress status as a proxy for further long-term harm in healthy subjects, using the well-established and fit-to-purpose measures of WBC and 8-epi-PGF2α, respectively, as indicators of the status of these pathways.

The study aims also at demonstrating additional benefits on other mechanistic pathways along with inflammation and oxidative stress by the means of additional biomarkers of potential harm (BoPH) and to assess association with functional benefits that are expected to be responsive to the extent of exposure to harmful and potentially harmful constituents (HPHCs).

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to understand the information provided in the main ICF and has signed the main ICF.
* Subject is 30-60 years old.
* Subject is healthy based on ECG, spirometry, vital signs, physical examination, medical history and Investigator's assessment.

Cigarette smokers:

* Has smoked ≥ 10 cigarettes/day on average (no brand restriction) over the past 2 years prior to screening.
* Has smoked ≥ 10 cigarettes/day on average (no brand restriction) for at least 10 years.
* Has not used other tobacco and nicotine products apart from cigarettes on a daily basis over the past 2 years prior to screening.
* Smoking status will be verified by urinary cotinine test (≥ 200 ng/mL) and CO breath test (≥ 10 ppm (1)).

THS users:

* Has used ≥ 10 HeatSticks/day on average over the past 2 years prior to screening.
* Has smoked ≥ 10 cigarettes/day on average (no brand restriction) for at least 8 years prior to switching to THS.
* Has smoked < 30 cigarettes/month and used other tobacco products or e-cigarettes < daily over the past 2 years prior to screening.
* Product use will be verified by urinary cotinine test (≥ 200 ng/mL) and CO breath test (< 10 ppm).

Former cigarette smokers:

* Has not smoked cigarettes or used any tobacco or nicotine-containing products on a daily basis over the past 2 years prior to screening.
* Has smoked ≥ 10 cigarettes/day on average (no brand restriction) for at least 8 years prior to stopping smoking.
* Smoking status will be verified by urinary cotinine test (< 100 ng/mL) and CO breath test (< 10 ppm).

Exclusion Criteria:

* As per the judgment of the Investigator, the subject cannot participate in the study for any reason (e.g., medical, psychiatric and/or social reason). The Investigator should specifically evaluate the subject's eligibility considering COVID-19 risk factors and local situation.
* The subject is legally incompetent or physically/mentally incapable of giving consent (e.g., emergency situation, under guardianship, in a social or sanitary establishment, prisoner or involuntarily incarcerated).
* The subject has/had clinically relevant diseases (including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrine, oncological, urological, immunological, pulmonary, and cardiovascular disease) or conditions that in the opinion of the investigator would jeopardize the safety of the subject or affect the validity of the study results.
* The subject has abnormal findings on physical examination, ECG, vital signs, spirometry or in the medical history, deemed clinically significant by investigators.
* The subject has/had within 30 days prior to screening a body temperature >37.5°C or an acute illness (e.g., upper-respiratory-tract infection, viral infection, etc.…) or the subject is confirmed or suspected active COVID-19 infection (based on the signs and symptoms observed at the time of assessment) at screening.
* The subject has used any prescribed or over-the-counter systemic medication with an impact on WBC or 8-epi-PGF2α within 5 half-lives of the medication prior to enrollment in the study (please refer to Appendix B).
* Subject has high blood pressure (hypertension), defined as > 139 mmHg systolic and/or > 89 mmHg diastolic or is currently treated with medication controlling high blood pressure.
* The subject has (FEV1/FVC) < 0.7 and FEV1 < 80% predicted value at post-bronchodilator (BD) spirometry.
* The subject has (FEV1/FVC) < 0.75 (pre-BD) and reversibility in FEV1 (that is both > 12% and > 200 mL from pre- to post-BD values).
* The subject has a history of allergic reactions to salbutamol.
* The subject has a body mass index (BMI) < 18.5 or ≥ 30 kg/m2.
* The subject has positive alcohol and/or drug screening test results.
* The subject has donated or received whole blood or blood products within 3 months prior to V1.
* The subject has been previously screened for this study.
* The subject is a current or former employee of the tobacco or e-cigarettes industry or of their first-degree relatives (parent, sibling, and child).
* The subject is an employee of the investigational site or any other parties involved in the study or of their first-degree relatives (parent, sibling, and child).
* The subject has participated in a clinical study within 3 months prior to V1.
* For women only: the subject is pregnant (does have a positive pregnancy test) or breast-feeding.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population was recruited through social media and traditional display advertising. The subjects included current cigarette smokers, current THS users (with a minimum of 2 years THS use), and former cigarette smokers (with a minimum of 2 years of smoking abstinence).
Sampling Method: Non-Probability Sample
Enrollment: 952 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Carboxyhemoglobin (COHb) in blood | Measured when subject visits study site on day 1.
  Carboxyhemoglobin (COHb) is assayed from whole blood. Expressed as % of saturation of hemoglobin.
Total 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (total NNAL) in urine | Measured when subject visits study site on day 1.
  Concentrations of total NNAL measured in urine and expressed as concentration adjusted for creatinine (pg/mg creat).
White Blood Cell total count (WBC) in blood | Measured when subject visits study site on day 1.
  Total count in blood (GI/L). Mean values are provided.
8-epi-Prostaglandin-F2α (8-epi-PGF2α) in urine | Measured when subject visits study site on day 1.
  Concentrations of 8-epi-PGF2α measured in urine and expressed as concentration adjusted for creatinine (pg/mg creat).

SECONDARY OUTCOMES:
High-Density Lipoprotein Cholesterol (HDL-C) | Measured when subject visits study site on day 1.
  Concentrations of HDL-C (mg/dL) measured in serum.
soluble Intercellular Adhesion Molecule-1 (sICAM-1) | Measured when subject visits study site on day 1.
  Concentrations of sICAM-1 (ng/mL) measured in serum.
11-dehydrothromboxane B2 (11-DTX-B2) | Measured when subject visits study site on day 1.
  Concentrations of 11-DTX-B2 measured in urine and expressed as concentration adjusted for creatinine (pg/mg creat).
Augmentation Index (AIx) | Measured when subject visits study site on day 1.
  The augmentation index (AIx) is a measure of systemic arterial stiffness, and is defined as the ratio of augmentation (Δ P) to central pulse pressure and expressed as percent. AIx = (ΔP/PP) x 100, where P = pressure and PP = Pulse Pressure.
Forced Expiratory Volume in 1 second (FEV1) %predicted, post-bronchodilator (post-BD) | Measured when subject visits study site on day 1.
  FEV1 post-bronchodilator and expressed as percentage predicted (FEV1 %pred).

OTHER OUTCOMES:
Neutrophil to Lymphocyte Ratio (NLR) | Measured when subject visits study site on day 1.
  Calculated by dividing the number of neutrophils by number of lymphocytes from serum.
High-sensitivity C-Reactive Protein (hs-CRP) | Measured when subject visits study site on day 1.
  Concentrations of hs-CRP (mg/dL) measured in serum.
Homocysteine (HCY) | Measured when subject visits study site on day 1.
  Concentrations of HCY (μmol/L) measured in plasma.
Myeloperoxidase (MPO) | Measured when subject visits study site on day 1.
  Concentrations of MPO (μg/L) measured in serum.
Triglycerides (TG) | Measured when subject visits study site on day 1.
  Concentrations of TG (mg/dL) measured in blood.
Fibrinogen | Measured when subject visits study site on day 1.
  Concentrations of Fibrinogen (mg/dL) measured in serum.
Glycated Hemoglobin (HbA1c) | Measured when subject visits study site on day 1.
  HbA1c measured in whole blood (%).
Forced Expiratory Volume in 1 second/Forced Vital Capacity (FEV1/FVC) ratio | Measured when subject visits study site on day 1.
  Measured with and without bronchodilator, absolute and % predicted values, where applicable.
Nicotine Equivalents (NEQ) in urine (expressed as concentration adjusted to creatinine) | Measured when subject visits study site on day 1.
  NEQ measured in urine and expressed as concentration adjusted for creatinine.
2-Cyanoethyl Mercapturic Acid N-Acetyl-S-(2-cyanoethyl)-L-cysteine (2CyEMA) | Measured when subject visits study site on day 1.
  2CyEMA measured in urine and expressed as concentration adjusted to creatinine.

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Haziza, PhD, Study Chair — Philip Morris Products S.A.
Locations (37):
- Bulgaria (4):
  - Medical Centre Asklepii, Kyustendil
  - Medical Centre Leo Clinic EOOD, Lovech
  - Medical Center ReSpiro, Razgrad
  - Medical Center Zara-Med EOOD, Stara Zagora
- Czechia (7):
  - Private Internal ambulance, Karlovy Vary
  - PreventaMed s.r.o., Olomouc
  - Praglandia s.r.o., Prague
  - Clintrial s.r.o., Prague
  - Zdravi - fit, s.r.o., Protivín
  - Ordinance praktickeho lekai'e, Přeštice
  - Vestra Clinics s.r.o., Rychnov nad Kněžnou
- Germany (11):
  - Velocity Clinical Research Germany GmbH, Berlin
  - emovis GmbH, Berlin
  - Synexus Clinical Research GmbH, Frankfurt
  - Klinische Forschung Hamburg GmbH, Hamburg
  - Klinische Forschung Hannover-Mitte GmbH, Hanover
  - Klinische Forschung Karlsruhe GmbH, Karlsruhe
  - Velocity Clinical Research Leipzig, Leipzig
  - Centrum für Diagnostik und Gesundheit, Klinische Forschung und Entwicklung, München
  - Schaum/Hecht_RED Institut fur medizinische Forschung und Fortbildung GmbH, Oldenburg in Holstein
  - Praxis Reinfeld Mitte, Reinfeld
  - Klinische Forschung Dresden GmbH, Sachsen
- Greece (2):
  - National and Kapodistrian University of Athens, Medical school, Attikon Hospital, 2nd Cardiology Department, Athens
  - Aristotle University Thessaloniki/Papageorgiou Hospital, Thessaloniki
- Japan (8):
  - Hakata Clinic, Fukuoka
  - Yokohama Minoru Clinic, Kanagawa
  - Nishikumamoto Hospital, Minami
  - OPHAC Hospital, Osaka
  - OCROM Clinic, Osaka
  - ToCROM Clinic, Tokyo
  - Samoncho Clinic, Tokyo
  - Sumida Hospital, Tokyo
- Poland (5):
  - Centrum Medyczne Pratia, Katowice
  - Clinical Medical Research Sp. z o.o., Katowice
  - Tomed Tomasz Miszalski-Jamka, Krakow
  - Synexus Polska Sp zoo OddziaL w Lodzi, Lodz
  - Bioresearch Group, Nadarzyn

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ansari SM, Leroy P, de La Bourdonnaye G, Pouly S, Reese L, Haziza C. Differences in biomarkers of potential harm after 2+ years of tobacco heating system use compared to cigarette smoking: a cross-sectional study. Biomarkers. 2025 Mar;30(2):178-191. doi: 10.1080/1354750X.2025.2461069. Epub 2025 Feb 19. PMID 39882959